CLINICAL TRIAL: NCT06630910
Title: New Technique of End to Side Two Layered and Stented Duct to Mucosa Pancreaticojejunostomy with Omental Wrapping During Whipple Operation
Brief Title: New Technique of Pancreaticojejunostomy During Whipple Operation
Acronym: whipple
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mahmoud Rady, MD, Lecturer of general surgery, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT (659)
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Periampullary Carcinoma Resectable; Pancreatic Tumors; Duodenal Neoplasms
Keywords: pancreaticoduodenectomy; omental flaps; whipple operation; periampullary neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Duodenal Neoplasms | interventions — Pancreaticojejunostomy; Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A double-layered, end-to-side pancreaticojejunostomy without stenting and omental patch (Active Comparator)
  Interventions: Procedure: Pancreaticojejunostomy without stenting and omental patch
- A double-layered, end-to-side pancreaticojejunostomy with stenting and omental patch (Active Comparator)
  Interventions: Procedure: Pancreaticojejunostomy with stenting and omental patch

INTERVENTIONS:
Procedure: Pancreaticojejunostomy without stenting and omental patch — A traditional pancreaticoduodenectomy with pylorus preservation was performed on each patient. A pancreaticojejunostomy was created by double-layered, end-to-side, duct-to-mucosa anastomosis between the primary pancreatic duct and jejunal wall without stenting or omental patch.
  Arms: A double-layered, end-to-side pancreaticojejunostomy without stenting and omental patch
Procedure: Pancreaticojejunostomy with stenting and omental patch — A traditional pancreaticoduodenectomy with pylorus preservation was performed on each patient. A pancreaticojejunostomy was created by double-layered, end-to-side, duct-to-mucosa anastomosis between the primary pancreatic duct and jejunal wall, a nelaton stent 6f was inserted into the pancreatic duct and jejunum of each patient receiving PJ. The larger omentum was separated longitudinally over an avascular zone, and one or two omental branches of the gastroepiploic arteries were preserved using pedicle omental flaps. The omental flap was pushed between the posterior surface of PJ and the portal vein, then wrapped over the anterior surface of PJ. The omentum was rolled up and secured with a few PDS sutures.
  Arms: A double-layered, end-to-side pancreaticojejunostomy with stenting and omental patch

SUMMARY:
Following pancreaticoduodenectomy, omental flaps around the pancreatic anastomosis can lower the risk of pancreatic fistula, post-pancreatectomy bleeding, and delayed gastric emptying. The overall morbidity following pancreaticoduodenectomy can be decreased with this straightforward and efficient treatment.

DETAILED DESCRIPTION:
A prospective analysis was conducted on the medical records of 48 patients who underwent pancreaticoduodenectomy at our institute for periampullary cancer between March 2022 and March 2024. A total of 24 patients who had undergone pancreaticoduodenectomy without a stent or omental wrapping around the pancreatic anastomotic site made up group A, while 24 patients who had undergone pancreaticoduodenectomy with a stent inside and omental wrapping made up group B. Patients with resectable tumors of the duodenum, ampulla, distal common bile duct, and pancreatic head met the inclusion criteria. Irresectability criteria (such as metastases, ascites, or arterial vascular invasion) were among the exclusion criteria.

A traditional pancreaticoduodenectomy with pylorus preservation was performed on each patient. Every patient had reconstruction utilizing a single jejunal loop after resection, which was made possible by various anastomoses. A pancreaticojejunostomy was created by double-layered, end-to-side, duct-to-mucosa anastomosis between the primary pancreatic duct and jejunal wall. The outer layer consisted of the residual pancreatic parenchyma and the seromuscular layer of the jejunum. An interrupted suture technique utilizing 4-0 monofilament polyglyconate was used to complete the pancreatic duct and jejunal mucosa anastomosis. A nelaton stent 6f was inserted into the pancreatic duct and jejunum of each patient receiving PJ. In group B, the larger omentum was separated longitudinally over an avascular zone, and one or two omental branches of the gastroepiploic arteries were preserved using pedicle omental flaps. The omental flap was pushed between the posterior surface of PJ and the portal vein, then wrapped over the anterior surface of PJ. The omentum was rolled up and secured with a few PDS sutures.

End-to-side hepaticojejunostomy was performed using interrupted sutures on the anterior wall and continuous 4-0 monofilament polyglyconate on the posterior wall. The gastrojejunal anastomosis was performed using a linear stapler. All patients underwent pancreatico-duodenectomy with a feeding jejunostomy tube placed 50 cm distal to the gastrojejunal anastomosis, using a silicone catheter 22f. Near drains are often seen panceraticojejunal and hepaticojejunal anastomoses. On the first postoperative day, the nasogastric tube was withdrawn, and all patients were started on FJ feeds on POD2 using the bolus approach, which involves administering the feeding solution 4-6 times a day, usually in 150-200ml sessions, over the course of 15-20 minutes, most frequently via a syringe. Once the patient was able to accept an oral diet, the FJ feed was discontinued. After three weeks of surgery, all FJ tubes were removed, and oral feeding was resumed as soon as the patient showed signs of improvement. The surgical process was the same in both groups, with the exception of omental wrapping and stenting, which were only done in group B. No patient got octreotide as a preventive measure. The institutional ethics committee gave its approval to the study. Follow up CT abdomen was done in all cases in group B to assess the pancreatic stent.

The following were the study's objectives: (a) On or after the third postoperative day, the drain outflow of any detectable volume was treated as a pancreatic fistula with an amylase content larger than three times the upper normal serum amylase value.] The pancreatic fistulae were graded according to ISGPF standards. According to surgical site infection (SSI) guidelines, (b) a high bilirubin content leak that lasted longer than five days and was observed in biliary fluid was classified as bile leakage; (c) an intra-abdominal abscess was diagnosed based on a culture-positive purulent collection and wound infection;(d) According to the International Study Group of Pancreatic Surgery (ISGPF) criteria, bleeding that happened within 24 hours of the index procedure was classified as early post-pancreatectomy hemorrhage, while bleeding that happened beyond that time was classified as late post-pancreatectomy hemorrhage; (e) The length of hospital stay was calculated as the day of surgery till the day of discharge from the hospital; (f) Postoperative mortality was the number of deaths that occurred within the hospital admission period or within 30 days after surgery; and (g) delayed gastric emptying was identified when the patient's nasogastric tube was left in place for three postoperative days, when the necessity for its reinsertion emerged after that day, or when the patient lost the ability to digest solid food after the seventh postoperative day.

Postoperative complications were categorized using the criteria established by Clavien and Dindo. The existence or lack of POPF was the main study's endpoint. The duration of hospital stay, the rate of complications overall, and the rate of surgical death were the secondary end goals.

ELIGIBILITY:
Inclusion Criteria:

Resectable tumors of the duodenum, ampulla, distal common bile duct, and pancreatic head.

Exclusion Criteria:

Irresectability criteria (such as metastases, ascites, or arterial vascular invasion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
The rate of pancreatic fistula after pancreaticoduodenectomy | 4 weeks postoperative
  On or after the third postoperative day, the drain outflow of any detectable volume was treated as a pancreatic fistula with an amylase content larger than three times the upper normal serum amylase value.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared upon request from the principle investigator.

REFERENCES:
- [Background] Ohwada S, Ogawa T, Kawate S, Koyama T, Yamada T, Yoshimura S, Sato Y, Tomizawa N, Ohya T, Morishita Y. Omentoplasty versus no omentoplasty for cervical esophagogastrostomy following radical esophagectomy. Hepatogastroenterology. 2002 Jan-Feb;49(43):181-4. PMID 11941948
- [Background] Smits FJ, Molenaar IQ, Besselink MG, Busch OR, van Eijck CH, van Santvoort HC; Dutch Pancreatic Cancer Group. Management of postoperative pancreatic fistula after pancreatoduodenectomy: high mortality after completion pancreatectomy: Reply to: Bressan et al. completion pancreatectomy in the acute management of pancreatic fistula after pancreaticoduodenectomy. HPB (Oxford). 2018 Dec;20(12):1223. doi: 10.1016/j.hpb.2018.05.015. Epub 2018 Jun 22. No abstract available. PMID 29941289
- [Background] Kolbeinsson HM, Chandana S, Wright GP, Chung M. Pancreatic Cancer: A Review of Current Treatment and Novel Therapies. J Invest Surg. 2023 Dec 31;36(1):2129884. doi: 10.1080/08941939.2022.2129884. Epub 2022 Oct 3. PMID 36191926
- [Background] Shah OJ, Bangri SA, Singh M, Lattoo RA, Bhat MY. Omental flaps reduces complications after pancreaticoduodenectomy. Hepatobiliary Pancreat Dis Int. 2015 Jun;14(3):313-9. doi: 10.1016/s1499-3872(15)60372-1. PMID 26063034
- [Background] Nikfarjam M, Kimchi ET, Gusani NJ, Shah SM, Sehmbey M, Shereef S, Staveley-O'Carroll KF. A reduction in delayed gastric emptying by classic pancreaticoduodenectomy with an antecolic gastrojejunal anastomosis and a retrogastric omental patch. J Gastrointest Surg. 2009 Sep;13(9):1674-82. doi: 10.1007/s11605-009-0944-1. Epub 2009 Jun 23. PMID 19548039
- [Background] Alverdy JC, Schardey HM. Anastomotic Leak: Toward an Understanding of Its Root Causes. J Gastrointest Surg. 2021 Nov;25(11):2966-2975. doi: 10.1007/s11605-021-05048-4. Epub 2021 Jun 7. PMID 34100248
- [Derived] Elmeligy HA, Azzam AM, Ossama Y, Rady M. New technique of end to side two layered and stented duct to mucosa pancreaticojejunostomy with omental wrapping during Whipple operation. BMC Surg. 2025 May 9;25(1):201. doi: 10.1186/s12893-025-02893-x. PMID 40346483